CLINICAL TRIAL: NCT06249412
Title: The Importance of Positive Expiratory Pressure Associated With the In-exsufflator in Patients With Amyotrophic Lateral Sclerosis on the Effectiveness of Therapy
Brief Title: The Importance of Positive Expiratory Pressure Associated With the In-exsufflator in ALS Patients
Acronym: PEPINEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Collaborators: French Physiotherapy Society / Société Français de Physiothérapie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A01269-36
Record Dates: First submitted 2024-01-26; First posted 2024-02-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis ALS7
Keywords: ALS; Amyotrophic Lateral Sclerosis; MI-E therapy; INEX therapy; Airway clearance technics; Neuromuscular disease; Cough assit
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis 7; Amyotrophic Lateral Sclerosis; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant (patient) will not see the treatment mode set on their INEX/MI-E. Only the care givers will know.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-E with Positive expiratory pressure during pause (PEP) (Experimental): With the MI-E EOVE-70 device, it is possible to enable the setting of PEP (Positive Expiratory Pressure) during the pause. When this setting is activated, PEP can be adjusted between 1 and 20 cmH2O. The MI-E session will last, depending on patient tolerance, between 8 and 15 minutes. In this study, the MI-E will be set in automatic or semi-automatic mode with settings proposed by the physiotherapists based on the effectiveness and tolerance of the patient. To titrate PEP, the practitioner will start at 8 cmH2O; the setting can be decreased or increased at the discretion of the practitioner to optimize it, based on the inspiratory volume and peak expiratory flow (PEF) measured by the device at each cycle (usual clinical practice). The practitioner can adjust PEP between a minimum of 4 and a maximum of 15 cmH2O. A wash-out period of 30 minutes is planned between each INEX session with and without the PEP function activated (Experimental arm and comparative arm)
  Interventions: Device: MI-E with PEP function activated during the pause
- MI-E without Positive expiratory pressure during pause (PEP) (Active Comparator): The MI-E session will last, depending on patient tolerance, between 8 and 15 minutes. In this study, the MI-E will be set in automatic or semi-automatic mode with settings proposed by the physiotherapists based on the effectiveness and tolerance of the patient. The PEP function will not be used by the practitioner (ie. 0 cmH2O of PEP during the pause). A wash-out period of 30 minutes is planned between each INEX session with and without the PEP function activated (Experimental arm and comparative arm)
  Interventions: Device: MI-E without PEP function activated during the pause

INTERVENTIONS:
Device: MI-E with PEP function activated during the pause — PEP function will be activated during the pause when using the EOVE-70. The PEP function in cmH2O will start at 8 cmH2O; the PEP setting can be decreased or increased at the discretion of the practitioner to optimize. The other therapeutic settings (positive pressure, negative pressure, inspiratory time, expiratory time and pause time) will be set individually for each patient by an experienced physiotherapist in order to reach the best clinical efficacy (usual clinical care)
  Arms: MI-E with Positive expiratory pressure during pause (PEP)
Device: MI-E without PEP function activated during the pause — The PEP function will not be activated during the pause when using the EOVE-70. The other therapeutic settings (positive pressure, negative pressure, inspiratory time, expiratory time and pause time) will be set individually for each patient by an experienced physiotherapist in order to reach the best clinical efficacy (usual clinical care)
  Arms: MI-E without Positive expiratory pressure during pause (PEP)

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a fatal neurodegenerative disorder that impairs motor neurons, with a life expectancy of 2 to 7 years after diagnosis. ALS manifests as 'spinal' when it primarily affects limbs, or 'bulbar' when it impairs speech and swallowing. The disease progressively weakens all skeletal muscles, causing respiratory issues and increased risk of lung infections due to ineffective coughing. Mechanical cough assistance via In-exsufflation therapy/ mechanical in-exsufflator devie (INEX/MI-E) applies positive and negative airway pressures non-invasively to improve coughing. However, MI-E may fail in some ALS patients due to airway collapse, often related to brainstem muscle dysfunction.Research by Andersen et al. in 2017 highlighted that during MI-E, ALS patients often experience adverse laryngeal movements, which can obstruct airways and reduce the therapy's effectiveness. To combat this, they suggested individualized MI-E settings to minimize airway collapse. Modern MI-E devices, such as the EOVE-70, offer adjustable positive expiratory pressure (PEP) between cycles to potentially enhance airway stability and coughing efficiency. The current study focuses on the impact of PEP during therapy pauses on the peak expiratory flow rate in ALS patients, which could lead to improved therapeutic outcomes.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is an incurable and debilitating neurodegenerative disease affecting both upper and lower motor neurons. The average life expectancy upon diagnosis ranges from 2 to 7 years. Treatment is symptomatic, aiming to manage symptoms rather than cure the disease. ALS can be classified as 'spinal' when symptoms primarily affect the limbs or 'bulbar' when the disease manifests with speech, swallowing, or coughing difficulties. Regardless of the subtype, ALS eventually affects all skeletal muscles, including respiratory muscles, leading to impaired coughing efficiency, secretion buildup, and increased lung infections. Enhancing cough efficiency is crucial for clearing airway secretions and reducing pneumonia risk.

In healthy individuals, coughing involves an increase in lung volume by inspiratory muscles, coordination of the glottis by laryngeal muscles, and increased thoracoabdominal pressure by expiratory muscles. This process is disrupted in ALS patients. In-exsufflation therapy is widely used and recommended to assist coughing mechanically by applying non-invasive positive and negative pressure changes through a mask. For MI-E to be effective and keep the upper airways open during therapy, coordinated glottic movements are essential. The ultimate goal is to increase peak expiratory flow (PEF) during coughing. However, in some patients, MI-E is ineffective due to the collapse of the upper airways during both phases of the therapy-insufflation and exsufflation-but especially during inspiration, possibly due to dysfunction of the muscles innervated by the brainstem.

In 2017, Andersen et al. demonstrated via laryngoscopies conducted during MI-E use that the therapy was associated with:

Adduction of the supraglottic laryngeal structures during the insufflation phase.

Retraction of the tongue base into the hypopharynx during insufflation. Adduction of the vocal cords in ALS patients during both insufflation and exsufflation, regardless of subtype.

These factors compromised the therapy's effectiveness, which aims to increase PEF during cough

Andersen et al. concluded that it is important to personalize and adjust the MI-E settings to reduce the risk of airway collapse and allow the maximum number of ALS patients to benefit from it.

Today, several MI-E devices are available on the market, sharing similar settings for target pressure (positive/negative), inspiratory/expiratory time, automation, etc. Notably, one particular device (EOVE-70, Eove, Pau) offers the use and adjustment of a positive expiratory pressure (PEP) during the pause (i.e., between each delivered cycle), which could reduce the risk of airway collapse during therapy, and improve cough expiratory flow rate as well as the tolerance and effectiveness of the treatment in ALS patients.

The aim of this study is to evaluate the effect of using the positive expiratory pressure function during the pause and before the following insufflation on the peak expiratory flow rate of cough in patients with ALS during MI-E therapy

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged over 18 years
* Patient with Amyotrophic Lateral Sclerosis (ALS)
* Patients with established or beginning bulbar disorders, identified by the healthcare team (speech impairment, hypersalivation, or swallowing difficulties)
* Patient naive to INEX therapy but prescribed for its installation or patient already treated by an INEX device
* Patient followed by the ALS mobile team of the Groupe Hospitalier du Havre or the CHU of Dijon
* Patient whose disease progression kinetics is medically deemed compatible with inclusion in the study
* Patient willing to participate in the research after receiving adequate information and the information letter.
* Patient affiliated with social security or a beneficiary of such a scheme.

Exclusion Criteria:

"● Patient not presenting an episode of infection or a past episode of respiratory infection less than one month old

* Mental illness interfering with the proper use of the device
* History of laryngospasm
* Inability to come for consultation with the ALS team of the Groupe Hospitalier du Havre or the CHU of Dijon
* Pregnancy
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure (patient under guardianship or curatorship) Article L1121-8.
* Appearance of a non-inclusion criterion
* Refusal to participate after inclusion
* Death from any cause"

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The average difference in PEF (Peak Expiratory Flow) in L/min with the use of the PEP function and without the use of this function. | Between 5 and 15 minutes (MI-E treatment period)
  We aim to study the effect of using PEP during the pause on cough peak expiratory flow (PEF) in patients with ALS during MI-E therapy. The PEF from all treatment cycles measured by an external pneumotachograph connected to the circuit between the machine and the patient will be averaged and compared between the arms: with and without PEP during the pause

SECONDARY OUTCOMES:
The average difference in inspiratory volume in mililiters with the use of the PEP function and without the use of this function. | Between 5 and 15 minutes (MI-E treatment period)
  We aim to study the effect of using PEP during the pause on inspiratory volume delivered in patients with ALS during MI-E therapy. The inspiratory volume from all treatment cycles measured by an external pneumotachograph connected to the circuit between the machine and the patient will be averaged and compared between the arms: with and without PEP during the pause
The perceived effect of PEP during pause on the effectiveness of MI-E therapy by the patient as well as their perceived comfort | Between 5 and 15 minutes (MI-E treatment period)
  We wish to measure the average difference on the VAS (Visual Analogue Scale) with the use of the PEP function and without the use of this function, for the sensation of effectiveness and comfort reported by the patient
Qualitative analysis of cough using flow/time graphs of patient coughs with the use of the PEP function and without the use of this function. | Between 5 and 15 minutes (MI-E treatment period)
  We wish to measure qualitatively (visually in post-analysis) the flow/time data recorded by the external pneumotachograph with the use of the PEP function and without the use of this function.
Comparison of PEF (Peak Expiratory Flow) reported by the MI-E machine versus PEF measured by the external pneumotachograph in L/min | Between 5 and 15 minutes (MI-E treatment period)
  We wish to compare the data reported by the device versus the data externaly recorded for a post-analysis comparison.
Comparison of Inspiratory Volume reported by the MI-E machine versus Inspiratory Volume measured by the external pneumotachograph in mililiters | Between 5 and 15 minutes (MI-E treatment period)
  We wish to compare the data reported by the device versus the data externaly recorded for a post-analysis comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- GH Havre, Le Havre, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided